CLINICAL TRIAL: NCT04758000
Title: Metformin as Maintenance Therapy in Patients With Bone Sarcoma and High Risk of Relapse
Acronym: Metform-Bone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Alessandra Longhi,MD, Medical Doctor, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 794/2020/Farm/IOR; 2020-002579-37 (EudraCT Number)
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Osteosarcoma; Ewing Sarcoma
Keywords: Metformin; poor responders osteosarcoma; post relapse bone sarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: 1. Group 1 Localized osteosarcoma that have presented a response ≤ 60% to the pre-operatory chemotherapy.
     Is expected the enrolment of 37 patients as total population, in 44 months. The patients will be followed for 3 years, started from the date of enrolment. Metformin will be administrated for 3 years maximum, unless there is a progression disease or if toxicity is verified.
  2. Group 2 Osteosarcoma and Ewing sarcoma patients with complete remission after the first relapse.
  Is expected the enrolment of 30 patients as total population, in 24 months. Metformin will be administrated at the Group 2 for 1 year. If there is no toxicity verified or relapse, the patient should continue the treatment for other 2 year (in a total 3 years as maximum).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): Metformin will be administrated according with patients body mass index (BMI). The study is divided into 2 groups.
  * Group 1: Localized osteosarcoma that have presented a response ≤ 60% to the pre-operatory chemotherapy).
  * Group 2: Osteosarcoma and Ewing sarcoma patients with complete remission after the first relapse.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin will be administrated according with patients body mass index (BMI).
  Patients between 14 and 18 years old or with BMI ≤ 20: 500 mg two times a day Patients older than 18 years or with BMI > 20: 850 mg two times a day.
  In all cases, metformin will be administrated for 3 years maximum, unless there is a progression disease or if toxicity is verified.

SUMMARY:
Primitive bone sarcoma are rare tumors with low options of therapy for patient treatment.

1. OSTEOSARCOMA VERY POOR RESPONDER COHORT. Necrosis on primitive localized osteosarcoma represents one of the principal prognostic factors. Nowadays, for localized osteosarcoma there is no maintenance therapy that have shown to be effective.

   In ISG-OS1 study in patients with necrosis < 60% had an event free survival (EFS) at 3 yrs of 20% (Ferrari S ) in a more recent analysis (Tsuda Y 2020) patients with a necrosis <60% had a 3 y EFS of 35% .
2. OSTEOSARCOMA AND EWING'S SARCOMA AFTER FIRST RELAPSE Maintenance therapy after Complete Remission occurring after Ewing's sarcoma or osteosarcoma patients is not a standard rule.

These patients when free from disease, after first relapse, are more likely to face a second relapse. EFS at ONE YEAR after first relapse in osteosarcoma is shown in literature to be around 21% (Leary SE 2013) and 16% (Tirtei E 2017). The EFS at ONE YEAR after first relapse in Ewing's sarcoma is inferior to 20% (Barker 2005, Ferrari S 2015). A maintenance therapy with low toxicity in these high risk patients could be an option.

Metformin has been reported to a reduce the incidence of different type of cancer in diabetic patients. Metformin is well tolerated in diabetics an it is used in other conditions in non diabetic, as ovarian polycystic syndrome, metabolic syndrome and obesity. Metformin has been employed as chemoprevention related to its mechanism of action in breast cancer (NCT01101438 ) and in pediatric cancer together with chemotherapy (NCT01528046).

This study aim to explore the effectiveness of metformin (a low cost and well tolerated drug) as maintenance therapy in osteosarcoma and Ewing sarcoma patients at high risk of relapse.

DETAILED DESCRIPTION:
MATERIALS & METHODS The study is divided in two groups

1. Group 1-Localized osteosarcoma that have reported a post neoadjuvant chemotherapy primary tumor necrosis ≤ 60% Metformin will be administrated for 3 years maximum or until progression disease or if G3 or G4 toxicity is verified.

37 patients as total population are necessary to evaluate a 3 yrs increase of EFS from 35% ( historical data Tsuda Y ) to 60%,

2. Group 2 Osteosarcoma and Ewing sarcoma patients in Complete Remission after the first relapse.Metformin will be administrated for 3 years or until progression .

The Event Free Survival of this second group will be calculated at 1 yr with the aim of an increase of EFS from 20%(historical data) to 45%

STATISTICAL ANALYSIS AND SAMPLE SIZE Sample size was calculated by the Expected Total Study Length minimization criteria to ensure a potency parameter of 80 % and point if there is a benefit in use Metformin compared to the historical control.

EFS will be estimated by Kaplan-Meier and the standard error will be used to calculate the interim analysis Z-factor as well as the final statistical analysis.

The final statistical analysis will be performed

* Group 1 after 3 years after last patient enrollment
* Group 2 at 1 year from the last patient enrollment : EFS at 1 year

OBJECTIVE

1. Evaluate the event free survival (EFS) in osteosarcoma and Ewing sarcoma patients with high risk of relapse compared to the historical control.
2. Evaluate Metformin's toxicity as maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Non metastatic osteosarcoma patients with necrosis ≤ 60 % in the end of post-operatory chemotherapy treatment (within 45 days.from the end of chemotherapy treatment).
* Osteosarcoma or Ewing sarcoma patients free from the disease after first relapse (within 45 days.from the local surgery or 45 days from the end of chemotherapy treatment).
* ≥ 14 years.
* Patient should not be participating in other clinical study.
* Patients should be able to swallow.
* Screening up to 30 days from the end of chemotherapy treatment or relapse.
* Start therapy up to 30 days from the screening.
* Normal renal function (creatinine <1,3 mg/L, clearance creatinine ≥ 70 ml/min) end liver function (total serum bilirubina <1,2 mg/dL, except Gilbert syndrome patients), AST e ALT <1,8 times the normal range value

Exclusion Criteria:

* Type B diabetic patient
* Metastatic patients
* Patients with acute metabolic acidosis (lactic acidosis, diabetic ketoacidosis).
* Patients with renal insufficiency (GFR < 70 ml/min).
* Patients with acute conditions that could cause kidney alterations as dehydration, severe infection and shock.
* Patients with hepatic insufficiency as acute alcohol intoxication and alcoholism.
* Patients with medical conditions that could cause tissue hypoxia: decompensated heart failure, respiratory failure, recent myocardial infarction, shock.
* Patient who does not meet the inclusion criteria
* Pregnant and breastfeeding patients, or young women at childbearing age who cannot exclude the state of pregnancy (possibly excluded by serum pregnancy test (BhCG test), in accordance with the recommendations of the CTFG.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 3 years
  Evaluate the event free survival (EFS) in osteosarcoma and Ewing sarcoma patients with high risk of relapse compared to the historical control

SECONDARY OUTCOMES:
Metformin toxicity | 3 years
  Evaluate Metformin's toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Longhi, MD, Principal Investigator — Istituto Ortopedico Rizzoli IRCSS, Bologna, Italy
Locations (1):
- Chemotherapy Div, Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Ferrari S, Bacci G, Picci P, Mercuri M, Briccoli A, Pinto D, Gasbarrini A, Tienghi A, Brach del Prever A. Long-term follow-up and post-relapse survival in patients with non-metastatic osteosarcoma of the extremity treated with neoadjuvant chemotherapy. Ann Oncol. 1997 Aug;8(8):765-71. doi: 10.1023/a:1008221713505. PMID 9332684
- [Background] Leary SE, Wozniak AW, Billups CA, Wu J, McPherson V, Neel MD, Rao BN, Daw NC. Survival of pediatric patients after relapsed osteosarcoma: the St. Jude Children's Research Hospital experience. Cancer. 2013 Jul 15;119(14):2645-53. doi: 10.1002/cncr.28111. Epub 2013 Apr 26. PMID 23625626
- [Background] Barker LM, Pendergrass TW, Sanders JE, Hawkins DS. Survival after recurrence of Ewing's sarcoma family of tumors. J Clin Oncol. 2005 Jul 1;23(19):4354-62. doi: 10.1200/JCO.2005.05.105. Epub 2005 Mar 21. PMID 15781881
- [Background] Ferrari S, Luksch R, Hall KS, Fagioli F, Prete A, Tamburini A, Tienghi A, DiGirolamo S, Paioli A, Abate ME, Podda M, Cammelli S, Eriksson M, Brach del Prever A. Post-relapse survival in patients with Ewing sarcoma. Pediatr Blood Cancer. 2015 Jun;62(6):994-9. doi: 10.1002/pbc.25388. Epub 2015 Jan 13. PMID 25585917
- [Background] Tsuda Y, Tsoi K, Parry MC, Stevenson JD, Fujiwara T, Sumathi V, Jeys LM. Impact of chemotherapy-induced necrosis on event-free and overall survival after preoperative MAP chemotherapy in patients with primary high-grade localized osteosarcoma. Bone Joint J. 2020 Jun;102-B(6):795-803. doi: 10.1302/0301-620X.102B6.BJJ-2019-1307.R1. PMID 32475245